CLINICAL TRIAL: NCT04272255
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of DPI-386 Nasal Gel Under Military Operational Conditions for the Prevention of Nausea Associated With Motion Sickness
Brief Title: Nasal Gel Under Military Operational Conditions for the Prevention of Nausea Associated With Motion Sickness
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DPI-386-MS-08
Record Dates: First submitted 2018-12-14; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DPI-386 nasal gel (Active Comparator): DPI-386 Nasal Gel is formulated to contain 0.2 mg scopolamine HBr per 0.1 g dose, with each dose therefore described as "0.2 mg / 0.1 g"
  Interventions: Drug: scopolamine HBr
- placebo nasal gel (Placebo Comparator): Placebo nasal gel product is the same but does not contain scopolamine HBr
  Interventions: Drug: scopolamine HBr
- Transderm Scop® (Experimental): TDS patch delivers 1.5 mg of scopolamine over a 72-hour period. TDS arm will apply two TDS patches over the six treatment days.
  Interventions: Drug: Transdermal Scopolamine

INTERVENTIONS:
Drug: scopolamine HBr — Nasal Gel
  Arms: DPI-386 nasal gel; placebo nasal gel
Drug: Transdermal Scopolamine — Patch
  Arms: Transderm Scop®

SUMMARY:
This multi-site Phase 3 clinical trial is a randomized, double-blind, placebo-controlled and open label active-controlled study to identify the safety and efficacy of a repeated-dose regimen of DPI-386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of motion sickness. The study will be conducted aboard Navy fleet or Marine ships undergoing military operations to obtain data in an operationally relevant real world environment.

DETAILED DESCRIPTION:
The study will have three arms: DPI-386 nasal gel, placebo nasal gel, and Transderm Scop® (1.5 mg/72 hours; transdermal scopolamine patch [TDS], the current standard of care for the treatment of motion sickness). The study will include 100 subjects per arm, for a total of 300 subjects (n=300). Multiple ships and ships' crews will be used, until the required enrollment is completed. The DPI-386 Nasal Gel and placebo nasal gel arms will be double-blinded, whereas the TDS arm will remain unblinded. Both DPI-386 Nasal Gel and placebo nasal gel will be administered twice daily over the six consecutive Treatment Days. The two daily doses of DPI-386 Nasal Gel or placebo nasal gel will be separated by a minimum of six hours ± 15 minutes, and will occur during the subject's on-duty period. The TDS patch will be administered on Treatment Days 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated ICD.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 to 59 (inclusive).
4. Active duty military or reserves on active status. All potential subjects must be able to provide a current military ID to be viewed by PI or qualified designee prior to signing the ICD.
5. At least minimally susceptible to provocative motion as evidenced by a minimum score of 3.0 on the Motion Sickness Susceptibility Questionnaire (MSSQ).
6. In good general health as evidenced by medical history with no recent history or current diagnosis of clinical problems as recommended by the PI or qualified designee.
7. Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.
8. For females of child-bearing potential: willingness to provide a urine sample for the hCG pregnancy test. Test must be negative.
9. Agreement to adhere to the following lifestyle compliance considerations:

   1. Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the six treatment days.
   2. Abstain from alcohol for 24 hours prior to first dose of study medication and during the six Treatment Days.

Exclusion Criteria:

1. Pregnancy, lactation, or positive urine pregnancy test at screening.
2. Known allergic reactions to scopolamine or other anticholinergics.
3. Currently prescribed any of the following medication types: belladonna alkaloids, antihistamines (including meclizine), tricyclic antidepressants, and muscle relaxants.
4. Hospitalization or significant surgery requiring hospital admittance within the past six months.
5. Treatment with another investigational drug or other intervention within the past 30 days.
6. Having donated blood or plasma or suffered significant blood loss within the past 30 days.
7. Having any of the following medical conditions within the last two years or deemed clinically significant by the PI or qualified designee as being exclusionary:

   1. Significant gastrointestinal disorder, asthma, or seizure disorders.
   2. History of vestibular disorders.
   3. History of narrow-angle glaucoma.
   4. History of urinary retention problems.
   5. History of alcohol or drug abuse.
   6. Nasal, nasal sinus, or nasal mucosa surgery.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of DPI-386 Nasal Gel | 3 days
  Compare the efficacy of DPI-386 Nasal Gel (0.2 mg scopolamine HBr per dose, maximum of two doses per day, for a maximum of six doses over three consecutive days) with that of the TDS patch and placebo nasal gel in the prevention and treatment of nausea associated with motion sickness. The efficacy endpoint will be determined by comparing the Motion Sickness Assessment Questionnaire (MSAQ) scores over the treatment period across all three treatment arm. Sixteen symptoms are listed, with symptoms differentiated along four dimensions: gastrointestinal, central, peripheral, and sopite-related. Each symptom is scored from 1 to 9 in severity and scores then calculated. All 16 items were collected from the general public instead of experts, allowing for a more accurate wording of the symptomology experienced by persons outside of hysiological sciences.
Safety of DPI-386 Nasal Gel in terms of cognitive effects | 24 hours
  Compare the safety of DPI-386 Nasal Gel with that of the TDS patch and placebo nasal gel, with an emphasis on cognitive effects by incidence of treatment related adverse events.

SECONDARY OUTCOMES:
Efficacy of DPI-386 and severe nausea | 3 days
  Compare the efficacies of DPI-386 Nasal Gel, TDS patch, and placebo nasal gel in severity of nausea. Respondents specify their degree of nausea by indicating a point along a continuous 100mm line between two end-points; left one is for "No nausea" and the right one for "Very severe nausea". Scoring is based on the length from left point and a higher score means more severe degree of nausea. Severity of nausea will measured by the Nausea Assessment (Visual Analog Scale) (VAS)) over the treatment period.
Safety of DPI-386 Nasal Gel in terms of cognition | 24 hours
  Compare the safety of DPI-386 Nasal Gel with that of TDS patch and placebo nasal gel in terms of cognition as measured by the Psychomotor Vigilance Tests (PVT). The (PVT) is a neurocognitive assessment that measures alertness and tests sustained attention and reaction time. It was originally developed for sleep studies, and involves simple reaction time testing by requiring the participant to push a button as soon as the stimulus (a light) appears. After a response, the reaction time (in ms) is displayed. The inter-stimulus interval varies from two to 10 seconds, so it is not predictable, and the entire task takes 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: David Helton, Study Director — Repurposed Therapuetics, Inc.
Locations (1):
- NAMRU-D, Dayton, Ohio, United States